CLINICAL TRIAL: NCT06164652
Title: Evaluation of the Validity of the Ceriter Stride One for Measuring Gait and Pressure Parameters in Healthy Adults
Brief Title: Evaluation of the Validity of the Ceriter Stride One in Measuring Gait and Pressure Parameters in Healthy Adults
Acronym: CSO-validity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2023-0104
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: comparing data (gait kinematics) gathered with GAITRite and Ceriter Stride One by walking at comfortable and increased speed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (M/V/X, 18-80) (Experimental)
  Interventions: Device: walking with Ceriter Stride One

INTERVENTIONS:
Device: walking with Ceriter Stride One — Subjects walk on the GAITRite with the CSO insole in their shoes.

SUMMARY:
The Ceriter Stride One is a certified medical device that aims to provide a better, more independent and safe gait pattern for people with neurological disorders, such as Parkinson's disease. The Stride One detects the (abnormal) gait pattern via an insole with pressure sensors and generates customised audio feedback (app), e.g. to avoid or correct Freezing or Gait (Parkinson's).

To gain more insight into the accuracy of the pressure and gait recordings, we want to compare them with those of the GAITRite. The GAITRite is an electronic walking carpet with an active zone 7.32m long and 0.61m wide. The carpet has pressure sensors embedded in horizontal lines. When a person steps on the carpet, these sensors capture the pressure distribution which, with the help of an algorithm, allows the collection of parameters per time unit (including speed, step time, stride time, cadence, etc.) and space (step and stride length, step and stride width, etc.). The GAITrite is considered a gold standard for capturing temporal and spatial data related to gait pattern.

Our research question can be answered by having healthy subjects step over the GAITRite with the Ceriter Stride One on, and then checking the agreement between spatiotemporal factors.

Thus, after IC and recording of administrative data, healthy adults will be invited for this cross-sectional validity study of a pressure-sensitive insole (Ceriter Stride One) against the validated and reliable gold standard, the GaitRite.

At intake, the informed consent is gone over and signed. The inclusion and exclusion criteria are then questioned in a short interview. Inclusion criteria are pain-free and safe walking. Exclusion criteria are pregnancy and (congenital or acquired) orthopaedic, neurological and other defects that make walking without a walking aid or orthosis (or shoe adaptation) painful, difficult and/or unsafe,

Ceriter insoles are placed in the test subjects' shoes, if possible in place of their own insoles, in case of orthotics on top. Via a Bluetooth transmitter, the captured signals from the pressure sensors are transmitted to and mobile phone and then via the internet to Ceriter's data portal where they are further processed and, for the purpose of this study, made available to the researchers.Subjects then step on the walking carpet with sensors (GAITRite) with these insoles in their shoes.Both systems record the pressures and analyse the gait pattern from there.

Each test subject is expected to step across the walking carpet at a comfortable pace for three full lengths and 3 lengths involving acceleration. This, fitted with the insoles, so that sufficient steps are available to average out step parameters.

The aim of the study is thus to find out to what extent the spatiotemporal parameters captured with the Ceriter Stride One coincide with those of the GaitRite.

DETAILED DESCRIPTION:
Results of previous research showed no statistically significant differences between the data from the insoles compared with those from the GAITrite.These insoles show promise for clinically assessing gait in individuals with Parkinson's disease as they offer the additional ability to collect continuous information over long periods of time and in real-world contexts.The insoles used involve a different type with different technical characteristics and provide additional opportunities for collecting continuous information over long periods of time and in real-world contexts.

The study will proceed as follows :

recruitment of 50 healthy adults. Appeal via flyer distributed via social media will publicise the study and appeal to voluntary interested parties.The flyer will state the inclusion criteria (healthy, 18-75, M/F/X) and exclusion criteria (being pregnant, not allowed/able to walk).

For interested people who contact us, the ICF will be explained and presented for signature before the corridor tests begin. Considered steps are :

(a) Give info to participant and check inclusion and exclusion criteria, sign IC b) Put on Ceriter Stride One device (place this sole in shoe, change with insole) - bilaterally c) walk over the Gaitrite (8m) with the following partims :

* standing (register pressure in stance) : ("stand on the line on the mat and stand still")
* start and step at a comfortable pace : 3 x ("step to the other side at a comfortable pace for you")
* start and accelerate (without walking) : 3x ("step to the other side, start slowly and gradually accelerate. While doing this, keep stepping, you do not have to run.") If the first attempt does not go well, a demonstration is given in addition to standardised instruction.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* M/V/X
* 18-80

Exclusion Criteria:

* pregnancy
* injuries/lesions which make walking painful or difficult

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
step length | 3 minutes
  n centimeter
step frequency / cadance | 3 minutes
  n steps per minute
gait speed | 3 minutes
  meter per second

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Cambier, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jacobs D, Farid L, Ferre S, Herraez K, Gracies JM, Hutin E. Evaluation of the Validity and Reliability of Connected Insoles to Measure Gait Parameters in Healthy Adults. Sensors (Basel). 2021 Sep 30;21(19):6543. doi: 10.3390/s21196543. PMID 34640868
- See also: The results showed no statistically significant differences between the data of the insoles compared to the data of the GAITRite. This means that the insoles are promising to assess clinically measurements of the gait pattern in pwPD. — https://pubmed.ncbi.nlm.nih.gov/34640868/